CLINICAL TRIAL: NCT02132143
Title: Comparative Study of Chemoradiation and Sequential Chemoradiation About Lung Adenocarcinoma Patients With Postoperative in pN2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hui Lin (Other)
Responsible Party: Sponsor-Investigator, Hui Lin, The president of the People's Hospital of Guangxi, People's Hospital of Guangxi Zhuang Autonomous Region
Organization: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LH-2014-XW
Record Dates: First submitted 2014-05-02; First posted 2014-05-07 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Lung Adenocarcinoma Patients With Postoperative in pN2
Keywords: Lung adenocarcinoma; Concurrent chemoradiotherapy; Sequential chemoradiotherapy; Progression-free survival
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progression-free survival&Concurrent chemoradiotherapy (Experimental): The first day of radiotherapy given pemetrexed(Powder for Injection) 500mg/m2 + cisplatin(Powder for Injection) 75mg/m2, two cycles of chemotherapy given during radiotherapy; then continue to give two cycles of consolidation chemotherapy, 21 days as a cycle.
  Intensity-modulated radiation therapy(IMRT),5000cGy～6000cGy/5～6W.
  Interventions: Radiation: intensity-modulated radiation
- Progression-free survival&sequential chemoradiotherapy (Active Comparator): Patients received adjuvant chemotherapy for four cycles,pemetrexed(Powder for Injection) 500mg/m2 + cisplatin(Powder for Injection) 75mg/m2, 21 days as a cycle.Then accept the Intensity-modulated radiation therapy(IMRT),5000cGy～6000cGy/5～6W.
  Interventions: Radiation: intensity-modulated radiation

INTERVENTIONS:
Radiation: intensity-modulated radiation — For concurrent chemoradiotherapy, the intensity-modulated radiation therapy(IMRT)will be given at the first day of therapy,total dose of 5000cGy～6000cGy/5-6 Weeks.
  Arms: Progression-free survival&Concurrent chemoradiotherapy
Radiation: intensity-modulated radiation — For sequential chemoradiotherapy,the intensity-modulated radiation will(IMRT) will be given when patients received adjuvant chemotherapy for four cycles,total dose of 5000cGy～6000cGy/5-6 Weeks.
  Arms: Progression-free survival&sequential chemoradiotherapy

SUMMARY:
The purpose of this study compares chemoradiation and sequential chemoradiation about Lung adenocarcinoma patients with postoperative in pN2 and then determines which therapeutic method is better for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Lung adenocarcinoma
* Postoperative staging pN2 period
* Voluntary participation and informed consent
* Age ≥ 18 years old, male or female, within six months of weight loss of less than 10%, can tolerate radiotherapy
* performance status( PS) score 0-2.
* Hemoglobin ≥ 80 g / L, white blood cell ≥ 4 × 109 / L, platelets ≥ 100 × 109 / L.
* Liver function: alanine aminotransferase (ALAT), aspartate transaminase (ASAT) <upper limit of normal (ULN) of 1.5 times, bilirubin <1.5 × ULN.
* Renal function: serum creatinine <1.5 × ULN.
* Compliance, and can be regular follow-up, voluntary compliance with study requirements

Exclusion Criteria:

* Do not meet the inclusion criteria
* There is evidence of distant metastases
* Suffered from other malignancies in five years
* Within the past January subjects received other drug trials
* Having serious allergies or idiosyncratic persons, such as you can not use folic acid, dexamethasone, vitamin B12 patients
* Severe lung or heart disease, a history
* Refuses or is unable to sign informed consent to participate in trials
* The abuse of drugs or alcohol addicts.
* Patients with difficult to control bacterial, viral, fungal infections
* Having a personality or mental disorders, without civil capacity or restricted civil capacity.
* Being pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | two and a half years
  01/01/2014-06/01/2016

SECONDARY OUTCOMES:
Overall survival | two and a half years
  01/01/2014-01/01-2016

OTHER OUTCOMES:
side-effect | one year
  06/01/2014-06/01/2015

CONTACTS AND LOCATIONS:
Locations (1):
- The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, China